CLINICAL TRIAL: NCT02492698
Title: Changes in Body Adiposity by Dual Probiotic Strains Positively Correlated With Changes in Lp-PLA2 Activity in Overweight Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LW_clinical
Record Dates: First submitted 2015-07-01; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Overweight
Keywords: Probiotic; Weight loss; Lp-PLA2
MeSH Terms: conditions — Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic group (Experimental): consumed 2 g of powder of a dual probiotic strains containing Lactobacillus curvatus HY7601 and Lactobacillus plantarum KY1032, twice a day after breakfast and dinner.
  Interventions: Dietary Supplement: Probiotic group
- Placebo group (Placebo Comparator): consumed 2g of powder that did not contain any probiotics, twice a day after breakfast and dinner.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Probiotic group — The 2 g of probiotic powder contained 0.1 g of Lactobacillus curvatus HY7601, 0.1 g of Lactobacillus plantarum KY1032, 1.24 g of crystalline cellulose, 0.5 g of lactose, and 0.06 g of blueberry-flavoring agent.
  Arms: Probiotic group
Dietary Supplement: Placebo group — The 2 g of placebo powder contained 1.34 g of crystalline cellulose, 0.6 g of lactose, and 0.06 g of blueberry-flavoring agent.
  Arms: Placebo group

SUMMARY:
The objective was to evaluate the effect of the consumption of dual probiotic strains containing Lactobacillus curvatus (L. curvatus) HY7601 and Lactobacillus plantarum (L. plantarum) KY1032 on weight loss, body adiposity and inflammatory markers including lipoprotein-associated phospholipase A2 (Lp-PLA2) activity in overweight subjects.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study was conducted on 120 subjects with age between 20 and 65 years, nondiabetic (fasting blood glucose <126 mg/dL and 2-hour blood glucose <200 mg/dL), and overweight (25 kg/m2 ≤ body mass index (BMI) < 30 kg/m2). Over a 12 week test period, the probiotic group consumed 2 g of powder twice a day containing L. curvatus HY7601 and L. plantarum KY1032, while the placebo group consumed the same product without probiotics for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65 years
* Nondiabetic (fasting blood glucose <126 mg/dL and 2-hour blood glucose <200 mg/dL)
* Overweight (25 kg/m2 ≤ body mass index (BMI) < 30 kg/m2)

Exclusion Criteria:

* Constant consumption of any probiotics products within 1 month before screening
* Unstable body weight (body weight change > 1 kg within 3 months before screening)
* Hypertension
* Type 2 diabetes
* Cardiovascular disease
* Cerebrovascular disease
* Thyroid disease
* Dietary supplementation within 6 months before screening
* Pregnancy or breast-feeding
* Medication affecting body weight, energy expenditure, glucose control or antibiotic treatment within 3 months before screening
* Acute or chronic infections
* Liver disease
* Kidney disease
* Gastrointestinal disease
* Cancer
* Medication or alcohol abuse
* Any other acute or chronic disease requiring treatment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Fat percentage by dual-energy x-ray absorptiometry (DEXA) at baseline and 12-week follow-up | 12-week follow-up
  Fat percentage (%)
Fat mass by DEXA at baseline and 12-week follow-up | 12-week follow-up
  Fat mass (g)
Lean body mass by DEXA at baseline and 12-week follow-up | 12-week follow-up
  Lean body mass (g)
Fat area by computed tomography (CT) at baseline and 12-week follow-up | 12-week follow-up
  Fat area (cm2) at levels of 1st lumbar (L1) vertebra and 4th lumbar (L4) vertebra

SECONDARY OUTCOMES:
Total Cholesterol at baseline and 12-week follow-up | 12-week follow-up
  Total Cholesterol (mg/dL)
HDL Cholesterol at baseline and 12-week follow-up | 12-week follow-up
  HDL Cholesterol (mg/dL)
LDL Cholesterol at baseline and 12-week follow-up | 12-week follow-up
  LDL Cholesterol (mg/dL)
Triglyceride at baseline and 12-week follow-up | 12-week follow-up
  Triglyceride (mg/dL)
High sensitivity C-reactive protein (hs-CRP) at baseline and 12-week follow-up | 12-week follow-up
  hs-CRP (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph.D., Principal Investigator — Dept. of Food and Nutrition, College of Human Ecology, Yonsei University, 50 Yonsei-ro, Seodaemun-gu, Seoul, 120-749, South Korea